CLINICAL TRIAL: NCT04611412
Title: Determination of Risk Factors for the Development of Obesity and Hypertension in Children According to Perinatal Programming of Metabolism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samarkand State Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Project #4
Record Dates: First submitted 2020-10-11; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; children; obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 group: Group I consisted of 17 people (16.83%) with a uniform type of obesity
  Interventions: Other: Risk Factors
- 2 group: Group II included 38 children with AO, and 20 of them had normal BLOOD pressure
  Interventions: Other: Risk Factors

INTERVENTIONS:
Other: Risk Factors — BMI in children and adolescents was compared with percentile charts developed by who for children from 5 to 19 years of age (WHO Growth Reference, 2007). Body mass index was defined as the ratio of body weight (in kg) to body length in the supine position or height in the standing position (m2).

SUMMARY:
to determine the risk factors for developing obesity in children with exogenous-constitutional obesity and arterial hypertension, according to the theories of early programming of metabolism

DETAILED DESCRIPTION:
A retrospective cohort study of 55 children aged 12 to 18 years (average 14.60±0.24 years) with exogenous-constitutional obesity was conducted, with 24 girls (43.6%) and 31 (56.4%) boys. Children were identified during dispensary examinations in family clinics in Samarkand in the period 2018-2019. All the examined children belonged to the Uzbek population.

ELIGIBILITY:
Inclusion Criteria:

* SDS (standart deviation score) of body mass index (BMI) ranging from +2.0 to +3.0

Exclusion Criteria:

* secondary obesity and overweight genetic syndromes,
* refusal of the child and/or parents to be examined

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: the cohort study will include 55 children aged 12 to 18 with exogenous constitutional obesity
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-02 (Estimated)

PRIMARY OUTCOMES:
Risk factors of metabolic syndrome | up to 36 months
  A retrospective, cohort study of 55 children aged 12 to 18 years with exogenous constitutional obesity will be conducted Children with exogenous-constitutional obesity were divided by the presence of abdominal (visceral) obesity and the presence of hypertension.
  Parents will be interviewed and medical records (forms 003/y and 112) of children with exogenous constitutional obesity will be analyzed. Also, on the basis of a specially developed questionnaire, children with exogenous constitutional obesity were surveyed. When conducting a survey of children and their parents, the following factors will be of particular importance: heredity, pregnancy, weight and body length at birth, the nature of nutrition in the first two years of life, eating habits, and physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Samarkand State Medical Institute, Samarkand, Uzbekistan

IPD SHARING:
Plan to Share IPD: No
Study participants will perform all types of medical and diagnostic activities